CLINICAL TRIAL: NCT00063375
Title: Interactive Computer Treatment for Panic Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Norman Schmidt, Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21MH062056 (NIH); R21MH062056 (NIH); DSIR AT-AS
Record Dates: First submitted 2003-06-25; First posted 2003-06-27 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Panic Disorder
MeSH Terms: conditions — Panic Disorder

INTERVENTIONS:
Behavioral: Computer Based Cognitive Behavioral Therapy

SUMMARY:
This study will develop an interactive computer-based version of cognitive behavioral therapy (CBT) and compare its effectiveness to book-based CBT for the treatment of panic disorder.

DETAILED DESCRIPTION:
Panic disorder (PD) is a highly prevalent and debilitating condition. Unfortunately, many people with PD go untreated because of the high cost and low availability of treatment. Research shows that CBT is an effective treatment for PD. When administered as a self-help, computer based treatment, CBT may provide a less expensive, more engaging treatment for PD.

Participants in this study will be randomly assigned to receive computer based treatment, book based treatment, or no treatment for 10 weeks. After these 10 weeks, symptoms of anxiety and depression will be measured with patient interviews, scales, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of panic disorder, with or without agoraphobia

Exclusion Criteria:

* Change in medication type or dose 12 weeks prior to study entry
* Suicidal
* Current substance abuse
* Current or past schizophrenia, bipolar disorder, or organic mental disorder. Patients on medications must meet stability requirements such that initial administration of the medication and dose has been maintained for at least 3 months prior to treatment and will be maintained until post-treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2002-01; Primary Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States